CLINICAL TRIAL: NCT07305753
Title: CanCan Body Composition Study
Acronym: Cancan
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Steven Heymsfield, Boyd Professor, Pennington Biomedical Research Center
Other Study IDs: PBRC 00006218
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants; Young Healthy Adults; Elderly (People Aged 65 or More)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-sectional group: 20 young (20-40yo) and 20 older (70+) adults

SUMMARY:
The aim of this study is to develop a dataset with reference body composition measurements using criterion methods. This dataset will be used to develop new protocols to study patients with cancer. Obtaining measurements of sodium bromide (NaBr), deuterium dilution (D2O), and D3-Creatine in a stratified sample of adults will determine the accuracy (and precision) of the available devices for ECW, TBW, and skeletal muscle mass measurements.

ELIGIBILITY:
Inclusion Criteria:

* Being either male or female
* Being an adult >20 - <40 or >70 years of age.
* Having a body weight of less than 440 pounds
* Being willing to comply with the study procedures
* Not having a chronic illness (e.g., diabetes, cancer, etc.)
* Must be willing to have biospecimens and imaging stored for research use

Exclusion Criteria:

* Being pregnant, attempting to become pregnant, or breastfeeding
* Having medical implants such as a pacemaker or metal joint replacements
* Having had a mastectomy, breast reduction, or breast implants
* Having hair that cannot fit in a swim cap
* Having a body weight greater than 440 pounds
* Taking medications that alter the body's fluid compartments (ex: diuretics)
* Not willing to have biospecimens and imaging stored for future research use.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be community dwelling, have a self-reported ability to walk one-quarter of a mile and climb 10 steps without difficulty, self-reported ability to perform activities of daily living (ADLs) without difficulty, and no life-threatening conditions or diseases that would alter their body composition from what is typical for their age, sex, and BMI. Overall, participants must be ambulatory, able to withstand lying flat on the DXA table for up to 10 minutes, stand without aid for 2 minutes, weigh less than 440 lbs and be in generally good health.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Mass | Single time point
  Muscle mass

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided